CLINICAL TRIAL: NCT04576039
Title: Ultrasonographic Appearance of the Endometrium After Saline Infusion in Women Presenting With a Thickened Endometrium After the Use of Ulipristalacetate.
Brief Title: Ultrasonographic Appearance of the Endometrium After Ulipristalacetate Use and Endometrial Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Stefan Cosyns, MD, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PAEC
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Uterine Fibroid; Endometrial Cyst
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- presenting with thickened endometruim (Experimental): women presenting with thickened endometrium after the use of ulipristalacetate will undergo a saline infusion in the uterus and immediate ultrasonographic control to visualise the morphology of the endometrium.
  Interventions: Diagnostic Test: saline infusion sonography

INTERVENTIONS:
Diagnostic Test: saline infusion sonography — Instillation of 10cc of saline infusion in the uterine cavity while performing an ultrasonic evaluation of the uterine cavity and endometrium.

SUMMARY:
If endometrial thickening is visualised (>10mm) after the use of ulipristalacetate in case of medical treatment for uterine fibroids a saline infusion and sonographic examination will be performed to evaluate the endometrium and exclude intra-uterine pathology.

DETAILED DESCRIPTION:
When ultrasonographic examination during follow up of a treatment with ulipristalacetate shows a thickening of the endometrium of 10mm or more ( thickening described in 10% of ulipristalacetate users and is completely benign), a saline infusion can help to exclude pathology in the uterine cavity. Saline infusion helps to better delineate the uterine cavity and endometrium. If fibroids or polyps are present in the uterine cavity they will clearly be seen.

This study was set up to describe how the endometrial changes after Esmya use appear on saline infusion sonography. This study can help to recognize ultrasonographic images in women presenting with thickened endometrium after Ulipristalacetate use.

ELIGIBILITY:
Inclusion Criteria:

* Women with thickened endometrium on ultrasound (defined as double endometrium thickness of ≥10mm) at the end of their treatment with ulipristalacetate.
* Normal double endometrium thickness before the use of ESMYA (<10mm)
* BMI >18 - < 30

Exclusion Criteria:

* Known type 0 or 1 fibroids
* Known intrauterine pathology

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
ultrasonographic morphology of the endometrium at saline infusion sonography | 1 week
  thickness and appearance of the endometrium

SECONDARY OUTCOMES:
diagnostic ability to exclude intrauterine pathology | 1week
  presence yes or no of intra uterine pathology as polyps or fibroids

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Degreef, PhD, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis UZBrussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No